CLINICAL TRIAL: NCT04176263
Title: The Impact of Split-belt Treadmill Training to Modulate Freezing-related Gait Deficits and Freezing Episodes in Parkinson's Disease
Brief Title: The Effect of Split-belt Treadmill Training on Gait in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S62825 (KUL); D454/13 (CAU); None was given (Other Grant/Funding Number: Jacques and Gloria Gossweiler Foundation)
Record Dates: First submitted 2019-11-16; First posted 2019-11-25 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease; Freezing of Gait
Keywords: Parkinson Disease; Freezing of Gait; Rehabilitation; Gait adaptation; Split-belt; Treadmill training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Overground turning speed during single and dual-task will be compared between a group who will receive 4 weeks of SBT 3 times a week and a group who will receive TBT in the same dose. Participants will be randomized (1:1) to either the SBT or TBT groups by an independent researcher who is not involved in the measurements of any of the studies using a computerized random number generation technique. The randomization will be stratified based on H&Y stage and freezing status (freezer/non-freezer).
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessors will be single blinded. Participants will be semi-blinded. The participants will be told that they can be assigned to one of the two forms of treadmill training.They do not know the exact content of the training they would receive and what training is given in the other arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBT (Experimental): The SBT group will receive a 4-week split-belt treadmill training program consisting of 3 training sessions every week. The training will have a progression of training duration over the four weeks. Participants will start at a total training duration of 30 minutes and this will be increased with 5 minutes every week. The maximal length will be 45 minutes of training. One session including breaks will take approximately 1 hour.
  Interventions: Behavioral: SBT
- TBT (Active Comparator): The TBT group will receive a 4-week tied-belt treadmill training program consisting of 3 training sessions every week. The training will have a progression of training duration over the four weeks. Participants will start at a total training duration of 30 minutes and this will be increased with 5 minutes every week. The maximal length will be 45 minutes of training. One session including breaks will take approximately 1 hour.
  Interventions: Behavioral: TBT

INTERVENTIONS:
Behavioral: SBT — The SBT group will receive a 4-week split-belt treadmill training, 3 times a week using a standardized progression protocol. The sessions, including breaks, will approximately take 1 hour each. The training will be given by a trainer experienced with PD.
  Arms: SBT
Behavioral: TBT — The TBT group will receive a 4-week tied-belt treadmill training, 3 times a week. To make sure exposure of the two interventions is similar the sessions of the TBT group will be of similar length and progression level (approximately 1 hour each). The training will be given by a trainer experienced with PD.
  Arms: TBT

SUMMARY:
People with Parkinson's disease (PD) often show gait impairments such as, shuffling gait, short steps and gait asymmetry and irregularity. These gait problems are already apparent in the early disease stages, having an immense effect on daily life functioning. Especially Freezing of Gait (FOG), where the patients are not able to initiate or continue their movement despite their intention to do so, is a debilitating problem. It is thought that lack of gait adaptability could be an underlying cause of FOG. With a split-belt treadmill the speed of both legs can be controlled independently, which forces participants to actively adapt their gait to the new situation. In a previous study performed at our lab, it was shown that only one session of split-belt training (SBT), in which the speed of one leg was reduced, improved gait adaptability and other gait features compared to tied-belt training (TBT). Furthermore, overground turning speed improved after only one single training session and this was even retained 24 hours later, indicating training induced long-term potentiation. Since the short-term effects of SBT are promising, the objective of this study is to investigate if 4 weeks of SBT, 3 times a week, has an effect on gait deficits found in individuals with PD, compared to 4-weeks, 3 times a week, of TBT.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of PD according to the recent criteria of the Movement Disorders Society made by a neurologist
2. Participants should be able to walk 5 minutes at a stretch without a walking aid
3. Hoehn & Yahr stage II or III in the ON state of medication
4. Mini Mental State Examination score of 24 or above
5. Participants should have a steady medication schedule at the start of the study (no change in the past month).
6. To be included as a freezer participant a score of at least 1 or higher should be recorded with the New Freezing of Gait Questionnaire.

Exclusion Criteria:

1. Current enrollment in another clinical study which may interfere with the conduction of this study.
2. Orthopedic injuries or other musculoskeletal problems, which could possibly effect balance and/or gait.
3. Unable or unwilling to commit to 4 weeks of training, 3 times a week
4. Participation in walking training in the month prior to the start of the study
5. Other neurological impairments (except PD)
6. Cardiovascular exercise risk factors diagnosed by a doctor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Average overground 360 degree turning speed (degrees/s) | Change in performance between the average overground turning speed from pre to post intervention (i.e. the week after the 4-week training period ended)
  Participants will be instructed to turn 360 degrees in alternating directions (clockwise/counterclockwise) for 60 seconds. The instruction is to turn as quickly as possible, while still feeling safe doing this. The average overground turning speed will be determined by the use of APDM Opal accelerometers which will be worn on both feet, wrists and the lower back.

SECONDARY OUTCOMES:
Average dual task overground 360 degree turning speed (degrees/sec) | Change in performance between the average overground turning speed from pre to post intervention (i.e. the week after the 4-week training period ended)
  Participants will be instructed to turn 360 degrees in alternating directions (clockwise/counterclockwise) for 60 seconds. The instruction is to turn as quickly as possible, while still feeling safe doing this. The average overground turning speed will be determined by the use of APDM Opal accelerometers which will be worn on both feet, wrists and the lower back. In addition to this task the participants also have to perform an auditory stroop task. The participant hears the words 'low' and 'high' in either a low or high pitch in random order and timing. The participant has to respond as quickly as possible to the pitch of the word and not to the word itself.
Retention of average overground 360 degree turning speed (degrees/sec) | Change in performance from post-intervention 1 week after the 4-week training period ended (Retest 1) to retention, 5 weeks later (Retest 2).
  Participants will be instructed to turn 360 degrees in alternating directions (clockwise/counterclockwise) for 60 seconds. The instruction is to turn as quickly as possible, while still feeling safe doing this. The average overground turning speed will be determined by the use of APDM Opal accelerometers which will be worn on both feet, wrists and the lower back.
Retention of dual task average overground 360 degree turning speed (degrees/sec) | Change in performance from post-intervention 1 week after the 4-week training period ended (Retest 1) to retention, 5 weeks later (Retest 2).
  Participants will be instructed to turn 360 degrees in alternating directions (clockwise/counterclockwise) for 60 seconds. The instruction is to turn as quickly as possible, while still feeling safe doing this. The average overground turning speed will be determined by the use of APDM Opal accelerometers which will be worn on both feet, wrists and the lower back. In addition to this task the participants also have to perform an auditory stroop task. The participant hears the words 'low' and 'high' in either a low or high pitch in random order and timing. The participant has to respond as quickly as possible to the pitch of the word and not to the word itself.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, PhD, Principal Investigator — KU Leuven; Christian Schlenstedt, PhD, Principal Investigator — Christian-Albrechts-University of Kiel
Locations (2):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium
- University Hospital Schleswig-Holstein (UKSH), Christian-Albrechts-University Kiel, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Seuthe J, D'Cruz N, Ginis P, Weisser B, Berg D, Deuschl G, Nieuwboer A, Schlenstedt C. Split-belt treadmill walking in patients with Parkinson's disease: A systematic review. Gait Posture. 2019 Mar;69:187-194. doi: 10.1016/j.gaitpost.2019.01.032. Epub 2019 Feb 7. PMID 30771729

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT04176263/SAP_000.pdf